CLINICAL TRIAL: NCT01065077
Title: A Placebo Controlled, Randomized, Double-Blind, Fixed-dose, Multicenter, Phase IIb Study to Investigate the Efficacy and Tolerability of BAY58-2667 (150 µg/h, 100 µg/h, 50 µg/h) Given Intravenously to Subjects With Acute Decompensated Chronic Congestive Heart Failure (ADHF)
Brief Title: BAY58-2667 Dose Finding Trial Investigating Fixed Doses in Patients With Acute Decompensated Chronic Congestive Heart Failure (ADHF)
Acronym: COMPOSE 1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14560; 2009-014377-40 (EudraCT Number)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2014-11

CONDITIONS: Acute Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — BAY 58-2667

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Cinaciguat (BAY58-2667)
- Arm 2 (Experimental)
  Interventions: Drug: Cinaciguat (BAY58-2667)
- Arm 3 (Experimental)
  Interventions: Drug: Cinaciguat (BAY58-2667)
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cinaciguat (BAY58-2667) — Infusion of 150 µg/h during 48h
  Arms: Arm 1
Drug: Cinaciguat (BAY58-2667) — Infusion of 100 µg/h during 48h
  Arms: Arm 2
Drug: Cinaciguat (BAY58-2667) — Infusion of 50 µg/h during 48h
  Arms: Arm 3
Drug: Placebo — Infusion of placebo during 48h
  Arms: Arm 4

SUMMARY:
A placebo controlled, double-blind and randomized study to assess different doses of a new drug (BAY58-2667) given intravenously, to evaluate if it is safe and can help to improve the well-being of patients with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-lactating female subjects, age >/= 18 years of age; or women without childbearing potential defined as postmenopausal women aged 55 years or older, women with bilateral tubal ligation, women with bilateral ovariectomy, and women with a hysterectomy
* Subjects must have the clinical diagnosis of CHF made at least three months prior to enrollment
* Subjects must experience worsening of both of the symptoms below leading to hospitalization at the time of entry into the study:

  * dyspnea and
  * clinical evidence of volume overload

Exclusion Criteria:

* Acute de-novo heart failure
* Acute myocardial infarction and/or myocardial infarction within 30 days
* Valvular heart disease requiring surgical intervention during the course of the study
* Heart failure due to or associated with uncorrected primary valvular disease, malfunctioning artificial heart valve, or uncorrected congenital heart disease
* Primary hypertrophic cardiomyopathy
* Acute inflammatory heart disease, eg, acute myocarditis
* Unstable angina requiring angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Pulmonary Capillary Wedge Pressure | 8 hours

SECONDARY OUTCOMES:
Cardiac index (CI) | 8 hours and 48 hours
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Follow up (30 + 5 days)
Right atrial pressure (RAP) | 8 hours and 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (55):
- United States (5):
  - Ridgewood, New Jersey
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Fairfield, Ohio
  - Philadelphia, Pennsylvania
- Austria (2):
  - Linz, Upper Austria
  - Vienna, Vienna
- Zagreb, Croatia
- Finland (2):
  - Helsinki
  - Oulu
- Germany (5):
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Homburg, Saarland
  - Erfurt, Thuringia
  - Jena, Thuringia
- Israel (3):
  - Haifa, Israel
  - Jerusalem, Israel
  - Tiberias, Israel
- Italy (5):
  - San Fermo della Battaglia, Como
  - Brescia
  - Ferrara
  - Mantova
  - Torino
- Japan (8):
  - Nagoya, Aichi-ken
  - Kure, Hiroshima
  - Higashiibaraki, Ibaraki
  - Kawasaki, Kanagawa
  - Ōmura, Nagasaki
  - Osaka, Osaka
  - Bunkyo-ku, Tokyo
  - Shinagawa, Tokyo
- Poland (6):
  - Gdansk
  - Lodz
  - Warsaw
  - Wroclaw
  - Zabrze
  - Zgorzelec
- Romania (2):
  - Bucharest
  - Cluj-Napoca
- Russia (2):
  - Krasnoyarsk
  - Moscow
- Serbia (3):
  - Belgrade
  - Kamenitz
  - Niš
- Slovakia (2):
  - Lučenec
  - Martin
- Slovenia (3):
  - Celje
  - Golnik
  - Ljubljana
- Sweden (2):
  - Gothenburg
  - Uppsala
- Switzerland (2):
  - Zurich, Canton of Zurich
  - Lugano, Canton Ticino
- Thailand (2):
  - Bangkok, Thailand
  - Bangkok

REFERENCES:
- [Result] Gheorghiade M, Greene SJ, Filippatos G, Erdmann E, Ferrari R, Levy PD, Maggioni A, Nowack C, Mebazaa A; COMPOSE Investigators and Coordinators. Cinaciguat, a soluble guanylate cyclase activator: results from the randomized, controlled, phase IIb COMPOSE programme in acute heart failure syndromes. Eur J Heart Fail. 2012 Sep;14(9):1056-66. doi: 10.1093/eurjhf/hfs093. Epub 2012 Jun 19. PMID 22713287
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/